CLINICAL TRIAL: NCT05867082
Title: Effects of Neural Mobilization on Respiratory Parameters, Pain, Range of Motion, and Neck Awareness in Patients With Chronic Neck Pain: A Randomized Controlled Trial
Brief Title: Effects of Neural Mobilization on Respiratory Parameters in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 009
Record Dates: First submitted 2023-05-09; First posted 2023-05-19 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain; Respiratory
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural Mobilization Group (Experimental): Each participant underwent 15 treatment sessions (5 days per week for 3 weeks). Further, in the NM group, in addition to conventional treatment, 10 sessions of neural mobilization were performed.
  Interventions: Other: Neural Mobilization
- Control Group (Experimental): Each participant underwent 15 treatment sessions (5 days per week for 3 weeks).
  Interventions: Other: Neural Mobilization

INTERVENTIONS:
Other: Neural Mobilization — Radial Nerve Mobilization, Medial Mobilization, Ulnar Mobilization

SUMMARY:
Objective: Neural mobilization (NM) is commonly used to treat nerve disorders, and it is useful for disorders associated with neck and arm pain. This study aimed to determine the effects of NM on respiratory function in patients with chronic neck pain.

Methods: Overall, 26 patients with neck pain were randomly assigned to two groups: NM or control. In these participants, respiratory function and active cervical range of motion were assessed before and after intervention. Furthermore, the participants were provided a visual analog scale (VAS) and Fremantle Neck Awareness Questionnaire (FreNAQ). Each participant underwent 15 treatment sessions (5 days per week for 3 weeks). Further, in the NM group, in addition to conventional treatment, 10 sessions of neural mobilization were performed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 25-65 years,
* those with neck pain for >3 months
* those with complaints of pain, tension
* numbness on neurodynamic nerve tests

Exclusion Criteria:

* individuals with spinal stenosis,
* neurological diagnosis, malignancy,
* upper extremity vascular problems,
* osteoporosis,
* pregnancy,
* history of newly repaired peripheral nerves,
* inflammatory processes,
* cervical spine and upper extremity surgeries,
* conditions affecting lung capacity (such as asthma, bronchitis, and diabetes mellitus)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test | Change from baseline respiratory function at 3 weeks
  PFTs were performed using a spirometer (Schiller SP-260). Spirometric measurements were obtained using a nasal clamp while the patient was in a sitting position. At least three measurements were obtained for each participant, and the best value was considered for the study. In PFT measurements, forced expiratory volume in the 1st second (FEV1), forced vital capacity (FVC), and FEV1/FVC values were compared between the two groups
Range of Motion (ROM) of the Joint | Change from baseline ROM at 3 weeks
  Participants' ROM of the neck was measured using a universal goniometer at baseline. The measurements for neck flexion, extension, lateral flexion, and rotation were made during active neck movements while the patient was in a seating position. For the measurement of ROM during neck flexion and extension, the goniometer was placed on the acromion, and the ROM was measured by following the midline of the ear. To measure ROM during lateral flexion, the goniometer was placed on the spinous process of the cervical vertebra 7, and the ROM was measured by tracking its movement. For the measurement of ROM during rotation, the goniometer was placed in the center of the head, and the ROM was measured by following the nose. All measurements were reported in degrees.
Pain Intensity | Change from baseline pain intensity at 3 weeks
  Pain intensity was assessed using Visual Analog Scale. A description of the parameter being evaluated was written at either end of a 10-cm horizontal line, with scores ranging from 0 (no pain) to 10 (excruciating pain). The participants were asked to choose the score that best described their pain

SECONDARY OUTCOMES:
Fremantle Neck Awareness Questionnaire (FreNAQ in Turkish (FreNAQ-T) | Change from baseline FreNAQ-T at 3 weeks
  FreNAQ-T is a Likert-type questionnaire that assesses individual-specific altered perception (0 = I never felt/never feel this way, 1 = I rarely feel this way, 2 = I sometimes or some of the time feel this way, 3 = I often feel this way, 4 = I always or most of the time feel this way). The questionnaire consists of nine questions, for example, about how they perceive their neck in relation to their body and how they perceive their body position. The total score ranges from 0 to 36. High score indicates a poor prognosis. Onan et al. (2020) developed the Turkish version of the questionnaire and assessed its validity and reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tunç, Msc, Study Director — Medical Park Gebze Hospital
Locations (1):
- Medical Park Gebze Hosptal, Gebze, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No